CLINICAL TRIAL: NCT02098018
Title: Comparison of Stress Reduction Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Principal Investigator, Sara W Lazar, Associate Research Scientist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R34AT007197 (NIH)
Record Dates: First submitted 2014-03-18; First posted 2014-03-27 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Program 1 (Active Comparator): Program 1
  Interventions: Behavioral: Program 1
- Program 2 (Active Comparator): Program 2
  Interventions: Behavioral: Program 2

INTERVENTIONS:
Behavioral: Program 2 — A well-established behavioral method for reducing stress. To maintain blinding, details will be given to participants after randomization.
  Arms: Program 2
Behavioral: Program 1 — A well-established behavioral method for reducing stress. To maintain blinding, details will be given to participants after randomization.
  Arms: Program 1

SUMMARY:
There are many ways to reduce stress. This study will compare 2 different programs for reducing stress. In addition to looking at how well the programs reduce stress, we will also ask questions about how these programs may be working.

ELIGIBILITY:
Inclusion Criteria:

* 25-50 years of age
* Able to engage in moderate physical activity
* Interested in being treated for stress

Exclusion Criteria:

* Use of psychotropic medications within 6 months prior to study.
* History of extreme physical or psychological trauma.
* Medical conditions that would interfere with study procedures or confound results, such as diabetes, pregnancy, or paralysis.
* Axis I psychiatric diagnosis; e.g., history of substance use disorder, psychotic disorder, bipolar disorder, or eating disorder.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress | baseline to 24 weeks
  Participants will complete a short questionnaire about how stressed they feel. There will be 4 time points: baseline, week 8, week 12, week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lazar, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - University of Connecticut- Storrs, Storrs, Connecticut
  - Massachusettts General Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Braun TD, Riley KE, Kunicki ZJ, Finkelstein-Fox L, Conboy LA, Park CL, Schifano E, Abrantes AM, Lazar SW. Internalized weight stigma and intuitive eating among stressed adults during a mindful yoga intervention: associations with changes in mindfulness and self-compassion. Health Psychol Behav Med. 2021 Nov 19;9(1):933-950. doi: 10.1080/21642850.2021.1992282. eCollection 2021. PMID 34868736